CLINICAL TRIAL: NCT03463109
Title: Locating Nociceptive Stimuli Applied to the Lumbar Region in Healthy Subjects and in Subjects With Chronic Low Back Pain
Brief Title: Locating Nociceptive Stimuli on Digital Body Chart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Alessandra Raschi, Principal Investigator, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Localizzazione Stimoli
Record Dates: First submitted 2018-02-22; First posted 2018-03-13 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Low Back Pain; Healthy Volunteers
Keywords: Chronic low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: The same procedure will be used for people with chronic low back pain and for healthy volunteers.
Who Masked: Participant
Masking Description: Every participant will recive stimulation on his back in a pre-defined random order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Other): Electrocutaneous stimulation. A standardized grid will be drawn over the participants' lumbar region. Circular electrodes, connected to a constant current stimulator, will be applied at points on the grid selected at random. Participants will be blinded to the electrode locations. Sets of painful electrocutaneous stimuli will be randomly delivered for each electrode. Participants will be instructed to draw with a stylus pen on a digital body chart displayed on a tablet the location on which they will perceive each painful stimulation.
  Interventions: Other: Electrocutaneous stimulation
- Chronic Low Back Pain (Other): Assessment + Electrocutaneous stimulation. Patients with chronic low back pain will be asked to provide information about their lifestyle, level of disability, current pain, general pain and to undergo an assessment of kinesiophobia and health status.
  After the assessment, a standardized grid will be drawn over the patients' lumbar region. Circular electrodes, connected to a constant current stimulator, will be applied at points on the grid. Patients will be blinded to the electrode locations. Sets of painful electrocutaneous stimuli will be randomly delivered for each electrode. Patients will be instructed to draw with a stylus pen on a digital body chart displayed on a tablet where they will perceive each painful stimulation.
  Interventions: Other: Assessment + Electrocutaneous stimulation

INTERVENTIONS:
Other: Electrocutaneous stimulation — Painful electrocutaneous stimuli will be randomly delivered to electrodes positioned in a random order on the participants' back. Participants will be instructed to draw with a stylus pen on a digital body chart displayed on a tablet where they will perceive each painful stimulation.
  Arms: Healthy Volunteers
Other: Assessment + Electrocutaneous stimulation — Patients will be asked to provide information about their lifestyle, level of disability, actual pain and general pain, assessment of kinesiophobia and health status.
  Subsequently, painful electrocutaneous stimuli will be randomly delivered to electrodes positioned in a random order on the patients' back. Patients will be instructed to draw with a stylus pen on a digital body chart displayed on a tablet where they will perceive each painful stimulation.
  Arms: Chronic Low Back Pain

SUMMARY:
Digital body charts are used to assess the pain experience in people with pain. People are asked to report their pain by shading a human body template on a digital tablet. The aim of this study is to investigate whether people with chronic low back pain, compared to healthy volunteers, consistently locate on a digital body chart all nociceptive stimuli induced in the lumbar region.

DETAILED DESCRIPTION:
Healthy volunteers and people presenting chronic low back pain, will be recruited. A standardized grid will be drawn over the participants' lumbar region. Circular electrodes, connected to a constant current stimulator, will be applied at points on the grid. All participants will be blinded to the electrode locations. Painful electrocutaneous stimuli will be randomly delivered for each electrode. Participants will be instructed to draw with a stylus pen on a digital body chart displayed on a tablet where they will perceive each painful stimulation.

The body chart will be centred on a canvas 768x1024 pixels (pxl), and pain location will be defined by X and Y coordinates. The consistency in reporting the location of each painful stimulation will be described through coordinates.

In addition, only people presenting chronic low back pain will be asked to provide information about their lifestyle, level of disability, actual pain and general pain, assessment of kinesiophobia and health status.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (duration more than three months)

Exclusion Criteria:

* denial of informed consent;
* presence of pacemaker;
* pregnancy or possible pregnancy status;
* lumbar surgery (spinal fusion);
* documented degenerative pathology of the central nervous system;
* documented concomitant pathology altering sensitivity (e.g. diabetes, fibromyalgia);
* reduced motor control of the dominant hand (reported by every subject as conditioning the writing and therefore the ability to compile the body chart);
* presence of skin moles and/or scars on the back that may interfere with the conduction of the electrical stimulus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
The distance from marked points to the representation of the stimulated point on the digital body chart. | Immediately after the electrocutaneous stimulation

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) score | Before electrocutaneous stimulation
  The Oswestry Disability Index is a tool for the assessment of a patient's functional disability. It is a self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.
  Each topic category is followed by six statements describing different scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5, where 0 indicates less amount of disability and 5 indicates most severe disability.
  The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
  Italian validated version of the scale will be used.
Current pain level on Visual Analogue Scale (VAS, 0-10 cm) | Before electrocutaneous stimulation
  The patient will be asked to draw a vertical line on a horizontal 10 cm line, where he/she felt the current pain intensity would be better represented, in a range from the left end of the line indicating "no pain" corresponding to 0 cm to the right one indicating "worst pain imaginable" corresponding to 10 cm.
  The total score of the scale ranges from 0 = "no pain" to 10 = "worst pain imaginable".
Recent pain (last week) level on Visual Analogue Scale (VAS, 0-10 cm) | Before electrocutaneous stimulation
  The patient will be asked to draw a vertical line on a horizontal 10 cm line, where he/she felt the recent pain intensity would be better represented, in a range from the left end of the line indicating "no pain" corresponding to 0 cm to the right one indicating "worst pain imaginable" corresponding to 10 cm.
Tampa Scale for Kinesiophobia (TSK-13) | Before electrocutaneous stimulation
  The Tampa Scale of Kinesiophobia (TSK) is a 13 item scale developed to measure the fear of movement (kinesiophobia) related to chronic lower back pain. Respondents are asked to rate each item on a 4-point Likert scale, ranging from 1 (strongly disagree) to 4 (strongly agree). The subscale ranges scores are 13-22 suggesting "subclinical level of kinesiophobia", 23-32 suggesting "mild level of kinesiophobia", 33-42 suggesting "moderate level of kinesiophobia" and 43-52 suggesting "severe level of kinesiophobia".
  Italian validated version of the scale will be used.
The Short Form Health Survey (SF-36) | Before electrocutaneous stimulation
  The Short Form Health Survey (SF-36) is a 36 item questionnaire which measures the quality of life across eight domains, which are both physically and emotionally based. High scores define a more favorable health state.
  Italian validated version of the scale will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Barbero, Study Director — University of Applied Sciences and Arts of Southern Switzerland
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all assessments (primary and secondary outcomes) will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Requestor will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Leoni D, Falla D, Heitz C, Capra G, Clijsen R, Egloff M, Cescon C, Baeyens JP, Barbero M. Test-retest Reliability in Reporting the Pain Induced by a Pain Provocation Test: Further Validation of a Novel Approach for Pain Drawing Acquisition and Analysis. Pain Pract. 2017 Feb;17(2):176-184. doi: 10.1111/papr.12429. Epub 2016 Mar 15. PMID 26992099
- [Result] Barbero M, Moresi F, Leoni D, Gatti R, Egloff M, Falla D. Test-retest reliability of pain extent and pain location using a novel method for pain drawing analysis. Eur J Pain. 2015 Sep;19(8):1129-38. doi: 10.1002/ejp.636. Epub 2015 Jan 6. PMID 25565607